CLINICAL TRIAL: NCT05696197
Title: Predicting Motor Learning of an Upper Limb Task Based on Behavioral and Disease-specific Characteristics in Patients With Parkinson's Disease
Brief Title: Learning Potential of Patients With Parkinson's Disease After Two Weeks of Targeted Touchscreen Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Alice Nieuwboer, Full Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S64842
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
Keywords: Neurological rehabilitation; Motor learning; Touchscreen skills; Home-based training
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Parallel, randomization in two groups (intervention/control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Practicing the Swipe Slide Pattern task in ST and DT conditions, offered in a random order over a period of 2 weeks, 5 days a week, approximately 10 minutes per training session. Training will be performed independently at home.
  Interventions: Behavioral: Targeted touchscreen training
- Control group (No Intervention): Participants in the control group will receive no intervention during the study period. They are given the opportunity to perform the SSP-training after the study period to ensure motivation in this group.

INTERVENTIONS:
Behavioral: Targeted touchscreen training — Participants will practice the Swipe Slide Pattern (SSP) task independently at home in both ST and DT condition, offered in a random order. During this task, participants form different pre-defined patterns by moving their finger over a touchscreen, resembling a touchscreen unlock trace. The DT condition includes the SSP-task while counting either red or green lights illuminated on the screen. They will receive 10 training sessions of the SSP-task over a period of two weeks. Each week will consist of 5 consecutive days of training for approximately 10 minutes per session. Participants will perform 9 trials of 12 patterns each, alternated with rest periods of 14 seconds. Instruction and answers are also included. Feedback will be provided by means of knowledge of performance. On each training day, participants will receive a reminder on the training tablet.
  Arms: Experimental group

SUMMARY:
Parkinson's disease (PD) is characterized by severe motor and non-motor symptoms, including upper limb dysfunction. Due to the degradation of dopaminergic neurons in the striatum, PD patients experience difficulties with motor learning and more specifically with the consolidation of motor memory. Recent work showed that intensive writing training improved writing skills in PD. Although consolidation effects were present, difficulties with retention were also still apparent. Besides impacting writing, manual dexterity deficits in PD can also affect the use of touchscreens. Researchers from our lab demonstrated that impairments were most pronounced in multi-direction sliding motions, indicating the need for training of these motor skills. Our lab demonstrated the classic difficulties with retention in PD after one session of training of a swipe and slide pattern on a tablet (SSP-task) as single task (ST), although immediate gains were demonstrated. Therefore, in this study the investigators will examine whether a two-week home-based training program of a tablet-based SSP-training program will lead to immediate and consolidated improvements that are retained in time. This program will combine ST and dual task (DT) training to provide variation during the training period, but also to increase the cognitive challenge during learning, thereby stimulation consolidation of learning. The primary aim of this study consists of investigating the learning effects after two weeks of targeted touchscreen training. Secondary, the investigators will examine whether these effects will also be retained after four weeks without practice and whether targeted training results in consolidated improvements, in terms of automaticity and transfer towards an untrained task. Given the objective recording of compliance to the training protocol, the investigators will explore the association between compliance rates and learning effects.

DETAILED DESCRIPTION:
Given the impaired touchscreen skills and the espoused difficulties with retention in PD, th e investigators will examine the training of touchscreen sliding motions delivered on a tablet enabling practice in the home setting. Both ST and DT conditions will be offered in a random order and feedback will be provided by means of knowledge of performance to enhance motivation and retention, as proved successful in previous work. The objective of this study is to examine the effects of this innovative training program immediately after two weeks of targeted training as the primary outcome in a randomized controlled trial (RCT). To resemble daily life as much as possible, all test and training sessions will be carried out in the ON-phase of the medication-cycle, i.e., approximately 1 hour after last medication intake. The effect of a 2-week home-based training program with a 4-week follow-up will be examined by including 36 PD patients, who will be randomized (strata: age, H&Y stage) in the experimental or control group. Sample size was based on the pilot study using the SSP-task showing an average movement time of 7.4s ± 3.43 in PD for sequence swiping at baseline in ST. Based on literature, the researchers assumed an improvement of 20.2% following training at retention. For the control group, the researchers expect a deterioration in performance of 5.6% after a period without training based on the changes observed in the control groups of recent studies investigating manual dexterity parameters over time. Using an α = 0.05 and β = 0.20, a sample size was calculated for repeated measures ANOVA analysis with a within-between factor interaction design (within: pre - post - retention; between: experimental group - control group). Consequently, total sample size was estimated at 30 participants. Taking a 20% dropout rate into account, this resulted in a total of 18 participants in each group.

The experimental group will train the SSP task for a duration of two weeks, whereas the control group will not receive any intervention. On day 1 (T0), all participants will undergo an extensive screening session, including motor and non-motor screening. Testing can be performed at the subject's home or in our laboratory according to patients' preference.

The average slide duration (in ms) and the accuracy (as the number of correctly formed patterns in %) on the SSP-task will be recorded as the main digitised outcomes, objectively recorded via the tablet. In addition to evaluating the immediate effects of touchscreen training, the investigators will also test retention effects after four weeks without training as a secondary outcome. Further, consolidation of learning will be assessed using secondary outcomes such as the SSP-test in ST and DT conditions to assess automaticity of learning, the mobile phone task to test transfer of learning (MPT, typing a predefined telephone number on a smartphone). As tertiary outcomes, specific questionnaires to capture motor and cognitive performance will be administered. Following the baseline session, the experimental group will receive 10 training sessions of the SSP-training (5 days/week, 10 min/session) over a period of two weeks. The training is home-based and unsupervised but is extensively explained by an expert trainer. The control group does not receive training. Both immediately after training (T1) and after a four-week retention period (T2), touchscreen motor skills will be re-assessed at home. The most appropriate linear mixed models will be used to analyse SSP performance, with group (intervention - control) as between-subject factor and time (baseline - post - retention) as within-subject factor. LEDD and other confounders will be included as covariates.

PD is a highly heterogeneous disorders, not only affecting motor but also cognitive functions. In fact, up to 80% of patients develops dementia over the disease course. Previous studies have identified global cognitive function as important determinants of training success. Therefore, cognitive function will be assessed extensively during the baseline session to investigate the association with training responsiveness. A global cognitive screen will consist of the Montreal Cognitive Assessment. Moreover, 2 specific tests will be used to assess each cognitive subdomain. Attention and working memory will be assessed using a digit and visual span forward and backward. The trail making test and alternating names test will be used for executive function. Visuospatial function will be examined using the short form of the Benton's judgement of line orientation and the Rey Osterrieth Complex figure. The 30-min recall of the latter test will also be used to assess memory, together with the Rey Auditory Verbal Learning test. The Boston naming test and the Animal fluency test of the Controlled Oral Word Association test will be used to assess language. Other non-motor features, such as anxiety, depression, and sleep quality, will be tested using validated questionnaires for PD.

Another important determinant of rehabilitation success is training compliance. However, previous studies have used self-reported logbooks of home-based exercise, which show high inter-participant variability. As such, our training program overcomes this limitation as training compliance is automatically recorded via the digitized training tablet. The investigators will explore whether compliance to training has an impact on learning effects within the training group by using a correlation analysis between compliance rates and training-related changes in performance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease based on the 'UK Brain Bank' criteria
* Hoehn and Yahr (H&Y) stage I-III, participants in H&Y stage I should have the right side as the most affected side
* Right handed, or right-handed use of touchscreen devices.

Exclusion Criteria:

* Cognitive decline (Mini Mental State Examination < 24)
* Comorbidities of the upper limb that could interfere with the study and are not caused by Parkinson's disease
* Other neurological disorders besides Parkinson's disease
* Color blindness as determined by the Ishihara test for color deficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Average slide duration (in ms) after two weeks of training | Baseline and post-training (2 weeks)
  The automatically recorded slide duration will be averaged and compared between the experimental group and the control group.

SECONDARY OUTCOMES:
Performance accuracy (in %) | Baseline, post (2 weeks) and retention (4 weeks)
  The performance accuracy will be calculated as the number of correctly performed patterns and will be compared between the experimental group and the control group.
Retention effects on average slide duration (in ms) after four weeks follow-up | Baseline, post (2 weeks) and retention (4 weeks)
  The automatically recorded slide duration will be averaged and compared between the experimental group and the control group.
Consolidation effects of two weeks of training | Baseline, post-training (2 weeks)
  Using the behavioral data gathered at the different time points described in Time frame, dual task interference will be calculated and compared between groups (experimental vs control), moreover the transfer towards an untrained task will be examined and compared between groups. The untrained task contains the mobile phone task, in which the time necessary to type in a predefined telephone number is recorded (in s).

CONTACTS AND LOCATIONS:
Overall Officials: Alice Nieuwboer, PhD, Principal Investigator — KU Leuven
Locations (1):
- Department of Rehabilitation Sciences KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nackaerts E, Heremans E, Vervoort G, Smits-Engelsman BC, Swinnen SP, Vandenberghe W, Bergmans B, Nieuwboer A. Relearning of Writing Skills in Parkinson's Disease After Intensive Amplitude Training. Mov Disord. 2016 Aug;31(8):1209-16. doi: 10.1002/mds.26565. Epub 2016 Mar 17. PMID 26990651
- [Background] Nieuwboer A, Rochester L, Muncks L, Swinnen SP. Motor learning in Parkinson's disease: limitations and potential for rehabilitation. Parkinsonism Relat Disord. 2009 Dec;15 Suppl 3:S53-8. doi: 10.1016/S1353-8020(09)70781-3. PMID 20083008
- [Background] Nackaerts E, Ginis P, Heremans E, Swinnen SP, Vandenberghe W, Nieuwboer A. Retention of touchscreen skills is compromised in Parkinson's disease. Behav Brain Res. 2020 Jan 27;378:112265. doi: 10.1016/j.bbr.2019.112265. Epub 2019 Sep 27. PMID 31568836
- [Background] Sidaway B, Ala B, Baughman K, Glidden J, Cowie S, Peabody A, Roundy D, Spaulding J, Stephens R, Wright DL. Contextual Interference Can Facilitate Motor Learning in Older Adults and in Individuals With Parkinson's Disease. J Mot Behav. 2016 Nov-Dec;48(6):509-518. doi: 10.1080/00222895.2016.1152221. Epub 2016 Jun 24. PMID 27340809
- [Background] Taghizadeh G, Azad A, Kashefi S, Fallah S, Daneshjoo F. The effect of sensory-motor training on hand and upper extremity sensory and motor function in patients with idiopathic Parkinson disease. J Hand Ther. 2018 Oct-Dec;31(4):486-493. doi: 10.1016/j.jht.2017.08.001. Epub 2017 Nov 14. PMID 29150384
- [Background] Correa TV, da Silva Rocha Paz T, Allodi S, de Britto VLS, Correa CL. Progressive muscle-strength protocol for the functionality of upper limbs and quality of life in individuals with Parkinson's disease: Pilot study. Complement Ther Med. 2020 Aug;52:102432. doi: 10.1016/j.ctim.2020.102432. Epub 2020 May 23. PMID 32951706
- [Background] Aarsland D, Andersen K, Larsen JP, Lolk A, Kragh-Sorensen P. Prevalence and characteristics of dementia in Parkinson disease: an 8-year prospective study. Arch Neurol. 2003 Mar;60(3):387-92. doi: 10.1001/archneur.60.3.387. PMID 12633150
- [Background] Lofgren N, Conradsson D, Joseph C, Leavy B, Hagstromer M, Franzen E. Factors Associated With Responsiveness to Gait and Balance Training in People With Parkinson Disease. J Neurol Phys Ther. 2019 Jan;43(1):42-49. doi: 10.1097/NPT.0000000000000246. PMID 30531385
- [Background] Strouwen C, Molenaar EALM, Munks L, Broeder S, Ginis P, Bloem BR, Nieuwboer A, Heremans E. Determinants of Dual-Task Training Effect Size in Parkinson Disease: Who Will Benefit Most? J Neurol Phys Ther. 2019 Jan;43(1):3-11. doi: 10.1097/NPT.0000000000000247. PMID 30531381
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] BLACKBURN HL, BENTON AL. Revised administration and scoring of the digit span test. J Consult Psychol. 1957 Apr;21(2):139-43. doi: 10.1037/h0047235. No abstract available. PMID 13416432
- [Background] Llinas-Regla J, Vilalta-Franch J, Lopez-Pousa S, Calvo-Perxas L, Torrents Rodas D, Garre-Olmo J. The Trail Making Test. Assessment. 2017 Mar;24(2):183-196. doi: 10.1177/1073191115602552. Epub 2016 Jul 28. PMID 26318386
- [Background] Hyde T, Fritsch T. Assessing executive function in Parkinson disease: the alternating names test. Part I. Reliability, validity, and normative data. Parkinsonism Relat Disord. 2011 Feb;17(2):100-5. doi: 10.1016/j.parkreldis.2010.08.023. Epub 2010 Nov 30. PMID 21123105
- [Background] Winegarden BJ, Yates BL, Moses JA, Benton AL, Faustman WO. Development of an optimally reliable short form for Judgment of Line Orientation. Clin Neuropsychol. 1998;12(3):311-314. doi:10.1076/clin.12.3.311.1992
- [Background] Gullett JM, Price CC, Nguyen P, Okun MS, Bauer RM, Bowers D. Reliability of three Benton Judgment of Line Orientation short forms in idiopathic Parkinson's disease. Clin Neuropsychol. 2013;27(7):1167-78. doi: 10.1080/13854046.2013.827744. Epub 2013 Aug 19. PMID 23957375
- [Background] Poreh A, Shye S. Examination of the Global and Local Features of the Rey Osterrieth Complex Figure Using Faceted Smallest Space Analysis Examination of the Global and Local Features of the Rey Osterrieth Complex Figure Using Faceted Smallest Space Analysis *. Clin Neuropsychol. 1998;12(4):453-467. doi:10.1076/clin.12.4.453.7240
- [Background] Schmidt M. Rey Auditory Verbal Learning Test: RAVLT : A Handbook. Western Psychological Services; 1996. https://books.google.be/books?id=UOcPRAAACAAJ
- [Background] Kaplan E, Goodglass H, Weintraub S. The Boston Naming Test. Lea & Fibiger; 1983.
- [Background] Tombaugh TN, Kozak J, Rees L. Normative data stratified by age and education for two measures of verbal fluency: FAS and animal naming. Arch Clin Neuropsychol. 1999 Feb;14(2):167-77. PMID 14590600
- [Background] Leentjens AF, Dujardin K, Pontone GM, Starkstein SE, Weintraub D, Martinez-Martin P. The Parkinson Anxiety Scale (PAS): development and validation of a new anxiety scale. Mov Disord. 2014 Jul;29(8):1035-43. doi: 10.1002/mds.25919. Epub 2014 May 23. PMID 24862344
- [Background] Almeida OP, Almeida SA. Short versions of the geriatric depression scale: a study of their validity for the diagnosis of a major depressive episode according to ICD-10 and DSM-IV. Int J Geriatr Psychiatry. 1999 Oct;14(10):858-65. doi: 10.1002/(sici)1099-1166(199910)14:103.0.co;2-8. PMID 10521885
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Schootemeijer S, van der Kolk NM, Ellis T, Mirelman A, Nieuwboer A, Nieuwhof F, Schwarzschild MA, de Vries NM, Bloem BR. Barriers and Motivators to Engage in Exercise for Persons with Parkinson's Disease. J Parkinsons Dis. 2020;10(4):1293-1299. doi: 10.3233/JPD-202247. PMID 32925106
- [Background] Schmidt M, Paul SS, Canning CG, Song J, Smith S, Love R, Allen NE. The accuracy of self-report logbooks of adherence to prescribed home-based exercise in Parkinson's disease. Disabil Rehabil. 2022 Apr;44(8):1260-1267. doi: 10.1080/09638288.2020.1800106. Epub 2020 Aug 7. PMID 32762573